CLINICAL TRIAL: NCT02816515
Title: Non Interventional Clinical Investigation of Ectoin® Mouth Wash for the Prevention and Treatment of Chemotherapy-induced Oral Mucositis
Brief Title: Ectoin® Mouth Wash for the Prevention and Treatment of Chemotherapy-induced Oral Mucositis
Status: Completed | Type: Observational
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016/EML/NIS
Record Dates: First submitted 2016-06-20; First posted 2016-06-28 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Mucositis
Keywords: Non interventional study; Ectoin; Mouth wash; Mucositis; Chemotherapy; Radiotherapy
MeSH Terms: conditions — Mucositis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Ectoin® mouth wash: The treatment will be started on the first day of radio- and/or chemotherapy, before development of mucositis
- Ectoin mouth wash: The treatment will be started after oral mucositis development in patients receiving radio- and/or chemotherapy
- Supersaturated electrolyte mouth rinse: The treatment will be started after oral mucositis development in patients receiving radio and/or chemotherapy

SUMMARY:
This is a 3-week, non-interventional, observational study of patients undergoing chemotherapy (sutent) designed as a three-arm parallel study. In this study, the efficacy of Ectoin containing mouthwash given prophylactically for the prevention of mucositis in patients before radio- and/or chemotherapy; as well as during radio- and/or chemotherapy for patients with mucositis compared to standard treatment should be investigated. The study doesn't intervene with routine treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving radio- and/or chemotherapy (sutent) and suffering from mucositis
* Female or male individuals ≥ 18 years

Exclusion Criteria:

* Male or female under 18 years
* Any disease that can, in the opinion of the treating physician, affect the outcome of the study
* Patients with known intolerance to one of the substances used
* Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with radio- and/or chemotherapy-induced mucositis
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2016-01; Primary Completion 2017-10-24 (Actual); Study Completion 2017-10-24 (Actual)

PRIMARY OUTCOMES:
Change in severity of oral mucositis as assessed by a visual examination and asking the patient about pain and discomfort | Visit 1(day 0), Visit 2(after 7 days), Visit 3 (after 14 days) and Visit 4 (after 21 days)
  A trained clinical member of the team scores the degree of oral mucositis, in accordance to the World Health Organization (WHO) mucositis scale as follow: grade 0, no signs or symptoms; grade 1, oral soreness and erythema; grade 2, oral erythema, ulcers and solid diet tolerated; grade 3, oral ulcers and liquid diet only; grade 4, oral alimentation impossible
Tolerability assessment of Ectoin Mouth Wash by using a subsequent patient questionnaire in the prevention and suppression of the severity of oral mucositis induced by radio- and/or chemotherapy. | day 21
Change in evaluation of pain on swallowing by using a patient-reported oral mucositis experience questionaire | Visit 1(day 0), Visit 2(after 7 days), Visit 3 (after 14 days) and Visit 4 (after 21 days)
  A patient-reported oral mucositis symptom score scale will be assessed to determine the severity of the symptom pain on swallowing over time on a 4-category scale ranging from 1 (none) to 4 (severe).
Change in evaluation of dry mucosa | Visit 1(day 0), Visit 2(after 7 days), Visit 3 (after 14 days) and Visit 4 (after 21 days)
  A patient-reported oral mucositis symptom score scale will be assessed to determine the severity of the symptom dry mucosa over time on a 4-category scale ranging from 1 (none) to 4 (severe).
Change in decreased saliva release | Visit 1(day 0), Visit 2(after 7 days), Visit 3 (after 14 days) and Visit 4 (after 21 days)
  A patient-reported oral mucositis symptom score scale will be assessed to determine the severity of the symptom decreased saliva release over time on a 4-category scale ranging from 1 (none) to 4 (severe).
Change in Irritation of mucosa | Visit 1(day 0), Visit 2(after 7 days), Visit 3 (after 14 days) and Visit 4 (after 21 days)
  A patient-reported oral mucositis symptom score scale will be assessed to determine the severity of the symptom irritation of mucosa over time on a 4-category scale ranging from 1 (none) to 4 (severe).
Change in swelling | Visit 1(day 0), Visit 2(after 7 days), Visit 3 (after 14 days) and Visit 4 (after 21 days)
  A patient-reported oral mucositis symptom score scale will be assessed to determine the severity of the symptom swelling over time on a 4-category scale ranging from 1 (none) to 4 (severe).

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by the Suspect Adverse Reaction Report Form (CIOMS Form I). | within 21 days after starting chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Lajos Géczi, PhD, Principal Investigator — National Institute of TB and Pulmonology
Locations (3):
- Hungary (3):
  - Department of Oncological Internal Medicine and Clinical Pharmacology "C", National Institute of Oncology Hungary, Budapest
  - National Koranyi Institute of TB and Pulmonology, Budapest
  - National Institute of Oncology, Department of Radiotherapy 7-9 Ráth György u., Budapest

REFERENCES:
- [Derived] Dao VA, Bilstein A, Overhagen S, Geczi L, Barath Z, Mosges R. Effectiveness, Tolerability, and Safety of Ectoine-Containing Mouthwash Versus Those of a Calcium Phosphate Mouthwash for the Treatment of Chemotherapy-Induced Oral Mucositis: A Prospective, Active-Controlled, Non-interventional Study. Oncol Ther. 2018 Jun;6(1):59-72. doi: 10.1007/s40487-018-0060-z. Epub 2018 May 9. PMID 32700140